CLINICAL TRIAL: NCT06573866
Title: Enhancement of Quality of Work And Life: A Personalised Primary Preventive Work Intervention to Enhance Sustainable Work Participation in Persons With Neurodegenerative Movement Disorders
Brief Title: Enhancement of Quality of Work And Life
Acronym: EQuAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); The Dutch Brain Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 115335
Record Dates: First submitted 2024-07-11; First posted 2024-08-27 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease; Hereditary Spastic Paraparesis; Cerebellar Ataxia; Mitochondrial Diseases; Neuromuscular Diseases (NMD)
Keywords: Neurodegenerative disorders; Work; Quality of life; Work-life balance; Randomized controlled trial; Need for recovery; Sustainable work participation; Preventive work intervention
MeSH Terms: conditions — Parkinson Disease; Spastic Paraplegia, Hereditary; Cerebellar Ataxia; Mitochondrial Diseases; Neuromuscular Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the PPWI (intervention) or the usual care (control) group, in a 1:1 ratio.
Masking Description: In the beginning of the trial, the investigator was masked. However, during the trial we decided that unmasking the investigator was more feasible, as the fully automatic procedures in Castor EDC eliminate the risk of influencing allocation or data collection for effectiveness outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preventive Participatory workplace intervention (PPWI) (Experimental): Participants in the PPWI group will receive the PPWI and continue to receive usual care.
  Interventions: Behavioral: Preventive Participatory workplace intervention
- Usual care control group (No Intervention): The usual care control group comprises usual care. There are no restrictions on usual care.

INTERVENTIONS:
Behavioral: Preventive Participatory workplace intervention — The Participatory Workplace Intervention (PPWI) is a process intervention in which a trained process facilitator guides an employee and their manager in identifying work-related obstacles or changes and finding solutions to overcome or manage these obstacles. Its primary goal is to achieve consensus between employee and manager with respect to the most obstructive obstacles for functioning at work and feasible solutions. Following consensus, the stakeholders formulate and agree upon a plan of action and execute the plan. In a subsequent meeting, the implementation of the plan of action will be evaluated. Six months after the evaluation, a follow-up will take place to determine whether new obstacles have emerged and whether a new cycle of process steps should be initiated.
  Arms: Preventive Participatory workplace intervention (PPWI)

SUMMARY:
Work participation is essential for quality of life, providing purpose, social interaction, financial security, and shaping social status. Work participation is increasingly compromised in people with slowly progressive chronic disorders (hereafter referred to as progressive disorders). This negatively impacts their quality of life. Early work-related support, focused on sustainable work-retention, has the potential to enhance work participation in people with progressive disorders. Therefore, this study investigates the (cost)effectiveness of the Preventive Participatory Workplace Intervention (PPWI), a personalized work intervention to enhance sustainable work participation. The investigators perform an 18-month randomized controlled trial (RCT). In addition, the investigators perform a process evaluation and an economic evaluation alongside the RCT. 124 Dutch working persons with three types of movement disorders will be included: Parkinson's Disease (PD), cerebellar ataxia (CA) and hereditary spastic paraparesis (HSP) and with slowly progressive neuromuscular and mitochondrial disorders.

DETAILED DESCRIPTION:
Work participation is essential for quality of life, providing purpose, social interaction, financial security, and shaping social status and personal identity. Work participation is increasingly compromised in people with progressive disorders. This negatively impacts their quality of life. People with slowly progressive chronic disorders (hereafter referred to as progressive disorders) lack (structural) work-related support. Early work-related support, focused on sustainable work-retention, has the potential to enhance work participation in people with progressive disorders. Therefore, the EQuAL-study (Enhancement of Quality of work And Life) investigates the (cost)effectiveness of the Preventive Participatory Workplace Intervention (PPWI), a personalized intervention to enhance sustainable work participation in people with progressive disorders. The aim of the study is to investigate study effects of the PPWI on need for recovery after work (primary endpoint), perceived self-efficacy at work, work-related well-being, quality of life and absenteeism (secondary outcomes). In addition, the PPWI's cost-effectiveness and cost-utility and its the process of implementation and mechanisms of impact will be explored (second and third aim, respectively). To address these aims, the investigators perform an 18 month randomized controlled trial (RCT). A cost and process evaluation will be performed alongside the RCT. 124 Dutch working persons with types of movement disorders will be included: Parkinson's Disease (PD), cerebellar ataxia (CA), and hereditary spastic paraparesis (HSP) and with slowly progressive neuromuscular and mitochondrial disorders. Participants will be recruited from approximately twelve regions across the Netherlands. Participants will be randomised to either the PPWI or an usual care control group in a 1:1 ratio. The PPWI is a process intervention in which a trained process facilitator guides an employee and their manager in identifying work-related obstacles or changes and finding solutions to overcome or manage these obstacles. Its primary goal is to achieve consensus between employee and manager with respect to the most obstructive obstacles for functioning at work and feasible solutions. There are no restrictions on usual care. The study will evaluate between-group differences from baseline to 18-month follow-up in need for recovery after work (primary endpoint) and self-efficacy at work and indicators of quality of life, work-related well-being, and productivity (i.e. absenteeism and presenteeism). For the second aim, the investigators will measure the costs associated with healthcare use, productivity loss, work-related adjustments, and the intervention. For the third aim, the investigators will evaluate the process in terms of implementation of the PPWI, its mechanisms of impact and the implementation context. The investigators envision the PPWI to support sustainable work retention while preserving work-life balance and quality of life for individuals with progressive disorders. Additionally, the trial will provide insights into which intervention components are effective and why. This will help potential future PPWI users in making informed decisions about whether the costs are justified by the anticipated value and benefits.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis Parkinson Disease, cerebellar ataxia, hereditairy spastic paraparesis, or a slowly progressive neuromuscular or mitochondrial disorder, confirmed by the treating physician (e.g. neurologist, rehabilitation physician)
* aged 18-65 years;
* being employed for at least 8 hours per week (at baseline). This also includes individuals who have reduced their working hours until reaching this threshold of 8 hours per week. Working time may be distributed across multiple working days;
* having the intention to continue to work during the study period of 18 months, to prevent inclusion of participants who plan to retire within the 18-month RCT period;
* being open to talk to the employer or manager about any changes or limitations in work performance (disclosing the diagnosis is not required, by law).

Exclusion Criteria:

* individuals who are at the beginning of a sick leave procedure (under the Gatekeeper Improvement Act; Wvp);
* being fully self-employed. Partial self-employment in addition to paid employment is allowed, on the condition that the paid employment accounts for more than half of the total weekly working hours;
* having a second employer for over eight hours per week;
* proficiency in the Dutch language is not sufficient;
* severe comorbidity or health-related event that will hamper compliance to the protocol, e.g. in case of a severe cognitive impairment, a relatively abrupt transition to a very progressive manifestation of the disease, a planned surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Need for recovery after work | Measured four times: at baseline, and after 6, 12 and 18 months
  Need for recovery after work is measured using the subscale need for recovery after work of the Dutch language version of the Questionnaire on the Experience and Evaluation of Work questionnaire (VBBA 2.0).

SECONDARY OUTCOMES:
Perceived self-efficacy at work | Measured four times: at baseline, and after 6, 12 and 18 months
  Perceived self-efficacy at work is measured with the self-efficacy at work scale. It measures one's perceived self-efficacy in solving work- and disease-related problems and consists of 14 5-point Likert scale items. A higher score indicates a higher level of self-efficacy.
Work home interference (WHI) | Measured four times: at baseline, and after 6, 12 and 18 months
  Work home interference (WHI) is measured with the subscale negative work-home interaction of the Survey Work-home Interaction - NijmeGen (SWING).
Limitations in work | Measured four timepoints: at baseline, and after 6, 12 and 18 months
  Limitations in work is measured with the Dutch language version of the Work Limitations Questionnaire (WLQ-mdlv).
Work-related stress | Measured four times: at baseline, and after 6, 12 and 18 months
  Work-related stress is measured with an 11-point single-item measure. The minimum value is 0 and maximum value is 10. A higher score indicates a higher level of experienced work-related stress.
Job satisfaction | Measured four times: at baseline, and after 6, 12 and 18 months
  Job satisfaction is measured wit an 7-point Likert scale single-item measure. The minimum value is 1 and maximum value is 7. A higher score indicates a higher level of job satisfaction.
Perceived balance in daily activities (i.e. life balance) | Measured four times: at baseline, and after 6, 12 and 18 months
  Percieved balance in daily activities as a parameter life balance, will be measured with the Dutch language version of the Occupational Balance Questionnaire (OBQ11-NL).
Health-related Quality of Life (QoL) | Measured four times: at baseline, and after 6, 12 and 18 months
  Health-related QoL is measured with the EuroQuality of Life Five Dimension (EuroQol 5D (EQ-5D-5L)).
Overall life satisfaction | Measured four times: at baseline, and after 6, 12 and 18 months
  Overall life satisfaction is measured with a single-item life satisfaction measure with an 11- point answer scale. The minimum value is 0 and maximum value is 10. A higher score indicates a higher level of life satisfaction.
Absenteeism | Measured four times: at baseline, and after 6, 12 and 18 months
  Absenteeism data include dates of sick and recovery notifications, working hours of absence, and whether the sick notification was related to the movement disorder. At the baseline measurement, absenteeism data will be collected through a questionnaire applying a recall period of three months. Upon participation, we ask participants to keep track of their absenteeism on a scheme we provide them with.
Presenteeism | Measured four times: at baseline, and after 6, 12 and 18 months
  Presenteeism refers to when employees show up to work despite being ill, that leads to reduced productivity. Presenteeism is measured with the presenteeism subscale of the iMTA Productivity Cost Questionnaire (iPCQ).

OTHER OUTCOMES:
Healthcare and occupational service utilization | Measured four three times: at 6, 12 and 18 months
  Primary and secondary healthcare and occupational service utilization (e.g. appointment with a rehabilitation physician, a physiotherapist or an occupational physician) will be measured through questionnaires. Participants will be asked to keep track of their healthcare and occupational service utilization over the past six months prior to each measurement. For this purpose, we provide participants with a scheme.
  Healthcare costs will be obtained by multiplying the utilization quantities with the costs per quantity, based on the cost calculation guidelines established for healthcare in the Netherlands in 2024. Occupational service utilization costs are calculated using tariffs for occupational service professionals.
Productivity (loss) costs (due to absenteeism) | Measured four times: at baseline, and after 6, 12 and 18 months
  Absenteeism data that are collected for the purpose of the effect evaluation, will be included as a third component.
  For the absenteeism costs, different calculation approaches will be used for the societal and employer's perspective (for the purpose of the economic evaluation). The societal perspective applies the iPCQ calculation guidelines, using the friction cost method. This method is based on the assumption that employees on long-term sick leave are eventually replaced. As a result, productivity losses primarily occur during the period required for an employer to replace an absent employee, known as the friction period. For the employer's perspective, absenteeism costs will be estimated using the Human Capital Approach (HCA).
Productivity (loss) costs (due to presenteeism and loss unpaid work) | Measured four times: at baseline, and after 6, 12 and 18 months
  Productivity loss due to presenteeism and loss unpaid work will be measured and valued using two iMTA Productivity Cost Questionnaire (iPCQ) modules [50], measuring productivity losses of paid work due to presenteeism and losses related to unpaid work. Costs will be calculated according to the iPCQ calculation guidelines and a standard production costs per hour.
Costs for work-related adjustments | Measured one timepoint: at 18 months
  Prior to T3, participants will be asked to retrieve data on work-related adjustments of the entire study period from their employer. The employer will be responsible for approving requested adjustments and must have documented the approval and any acquisition of the adjustments. Adjustments include material adjustments, such as an adapted desk chair, as well as adjustments like employing an assistant who takes over certain tasks. At T3, participants will fill in these requested data through a questionnaire.
  If costs for the adjustments are not provided together with the adjustment-data by the employer, average costs for acquisition of the adjustments will be used.
Intervention costs | After every intervention-session with a participant, from the date on which the first participant starts with the intervention until 18 months after the date of inclusion of the last participant.
  Data on time spent on the PPWI trajectory by process facilitators will be collected continuously through checklists. Process facilitators will report the actual (direct) time and indirect participant-related time spent per meeting, and, if applicable, the travel time. The intervention costs will be calculated by multiplying the hours registered by the process facilitators with the tariffs for occupational therapy in the Netherlands.
Recruitment (process evaluation outcome) | Pre-intervention (2 weeks before start recruitment),during recruitment period (monthly registration), 2 weeks after end recruitment period.
  Recruitment strategies that are used to reach and recruit participants. The recruitment strategies are registered by the investigator.
Reach (process evaluation outcome) | Weekly registration, from the date of randomization of the first participant until the date of randomization of the last participant, assessed up to 18 months.
  Proportion of the target audience that participates in the intervention. Reach is determined, based on: the number of individuals invited to participate in the trial, number of individuals potentially interested and the number of participants who participated (in the intervention group).
  Data on these variables are registered by the intervention providers.
Dose delivered (process evaluation outcome) | After every intervention-session with a participant, from the date on which the first participant starts with the intervention until 18 months after the date of inclusion of the last participant.
  Dose delivered is determined by the amount of meetings planned and intervention steps provided according to the protocol by the intervention providers. Dose delivered is determined, based on: the number of meetings that have taken place and the number of process steps that have been performed.
  Data on these variables will be retrieved from the intervention providers, by questionnaires.
Dose received (process evaluation outcome) | Post-intervention (at 18 months after baseline)
  Dose received is the extent to which participants actively engage with the intervention. Dose received is determined, based on: the extent to which all stakeholders involved have implemented the solutions as proposed during the participatory workplace intervention.
  Data on this outcome is retrieved by both participants and intervention providers, by questionnaires.
Fidelity (process evaluation outcome) | After every intervention-session with a participant, from the date on which the first participant starts with the intervention until 18 months after the date of inclusion of the last participant.
  Fidelity is the extent to which the intervention steps are delivered according to the protocol. Fidelity is determined, based on: whether the predefined fidelity criteria have been reached.
  Data on fidelity is retrieved from the intervention providers, by a questionnaire.
Quality of delivery (process evaluation outcome) | Post-intervention (at 18 months after baseline)
  Perceived quality of the delivery of the intervention by the intervention providers. Data on quality will be retrieved from participants, by a questionnaire.
Satisfaction with the intervention (process evaluation outcome) | Post-intervention (at 18 months after baseline)
  Satisfaction with the intervention in general, intervention steps, materials of the intervention, the intervention provider and the solutions that came out of the intervention.
  Data on satisfaction with the intervention will be retrieved from participants, by a questionnaire.
Perceived impact (process evaluation outcome) | Post-intervention (in period of 18-20 months after baseline)
  Perceived impact/effect is determined, based on: whether and how participants experienced that the intervention improved working and/or living conditions and functioning and which components of the intervention contributed to that (or not) Data on perceived impact of the intervention will be retrieved from (a subset of) participants, through semi-structured in-depth interviews.
Perceived benefit for participants (process evaluation outcome) | 1 year after inclusion of last participants
  Perceived benefit for participants is determined, based on: whether and how intervention providers perceived that the intervention improved working and/or living conditions and functioning of participants and which components of the intervention contributed to that (or not).
  Data on perceived benefit will be retrieved from the intervention providers, through focus-group interviews.
Facilitators and barriers (process evaluation outcome) | Post-intervention (in period of 18-20 months after baseline)
  Factors that either facilitate or hamper functioning and implementation of the intervention.
  Data will be retrieved from both intervention providers through focus-group interviews and from (a subset of) participants, through semi-structured in-depth interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Elbrich Postma, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Relevant and anonymised research data will be shared/published in the Radboud Data Repository (RDR) to guarantee long-term accessibility to the research data of the project of this research.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the measurements and analysis, relevant and anonymised research data will be placed on the RDR.
Access Criteria: The pseudonymized research data will be accessible in the RDR under restricted access. This means that researchers who are interested in re-use of the data are asked to contact the central contact person for permission. Approval is given after a signed agreement.